CLINICAL TRIAL: NCT01393743
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Adjunctive Perampanel in Primary Generalized Tonic Clonic Seizures
Brief Title: A Efficacy and Safety Study of Adjunctive Perampanel in Primary Generalized Tonic Clonic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2007-G000-332
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Seizure Disorder Generalized Tonic Clonic
Keywords: Central Nervous System
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Perampanel (Experimental): Participants received 6 tablets (initially 1 tablet of 2-mg perampanel plus 5 tablets of perampanel matched placebo) and up-titrated weekly in 2-mg increments to a target dose range of 8 mg per day maintaining the blind with administration of 6 tablets per day of either perampanel/placebo.
  Interventions: Drug: Perampanel
- Placebo (Placebo Comparator): Participants received 6 tablets of perampanel matched placebo, once a day.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Perampanel
  Other Names: E2007
  Arms: Perampanel
Drug: Placebo comparator
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy, safety, and pharmacokinetics (PK) of perampanel on Primary Generalized Tonic Clonic (PGTC) seizure frequency in adolescents and adults maintained on one to two stable antiepileptic drugs (AED).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, adjunctive-therapy study with an open-label Extension Phase. The Core Study consists of 2 phases: Prerandomization and Randomization. The Prerandomization Phase consisted of 2 periods: Screening (up to 4 weeks) and Baseline (4 or 8 weeks, depending on the accuracy of diary-documented seizures during Screening), during which participants will be assessed for eligibility to participate in the study. The Randomization Phase consisted of 3 periods: Titration (4 weeks), Maintenance (13 weeks), and Follow-up (4 weeks; only for those participants not entering into the Extension Phase). At the start of the Randomization Phase, eligible participants will be randomized to the perampanel or placebo treatment groups in a 1:1 ratio. The extension phase consists of 142 weeks.

ELIGIBILITY:
Inclusion:

1. Clinical diagnosis of PGTC seizures (with or without other subtypes of primary generalized seizures) and experiencing greater than or equal to 3 PGTC seizures during the 8-week period prior to randomization
2. Have had a routine electroencephalogram (EEG) prior to or during the Baseline Period with electroencephalographic features consistent with primary generalized epilepsy; other concomitant anomaly should be explained by adequate past medical history
3. On a fixed dose of one to a maximum of three concomitant antiepileptic drugs (AEDs) for a minimum of 30 days prior to Baseline; only one inducer AED (i.e., carbamazepine, oxcarbazepine, or phenytoin) out of the maximum of two AEDs will be allowed
4. A vagal nerve stimulator (VNS) will be allowed, but it must have been implanted greater than or equal to 5 months prior to Baseline (stimulator parameters cannot be changed for 30 days prior to Baseline and for the duration of the study).
5. Have had a computed tomography (CT) or magnetic resonance imaging (MRI) within the last 10 years (for adults) and 5 years (for adolescents) that ruled out a progressive cause of epilepsy
6. A ketogenic diet will be allowed as long as the participant has been on this diet for 5 weeks prior to randomization

Exclusion:

1. A history of status epilepticus that required hospitalization within 12 months prior to Baseline
2. Seizure clusters where individual seizures cannot be counted
3. A history of psychogenic seizures
4. Concomitant diagnosis of Partial Onset Seizures (POS)
5. Progressive neurological disease
6. Clinical diagnosis of Lennox-Gastaut syndrome
7. If felbamate is used as a concomitant AED, participants must be on felbamate for at least 2 years, with a stable dose for 60 days prior to Baseline. They must not have a history of white blood cell (WBC) count below less than or equal to 2500/microL (2.50 1E+09/L), platelets less than 100,000/microL, liver function tests (LFTs) greater than 3 times the upper limit of normal (ULN), or other indication of hepatic or bone marrow dysfunction while receiving felbamate.
8. Concomitant use of vigabatrin: Participants who took vigabatrin in the past must be discontinued for approximately 5 months prior to Baseline, and must have documentation showing no evidence of a vigabatrin-associated clinically significant abnormality in an automated visual perimetry test
9. Concomitant use of barbiturates (except for seizure control indication) within 30 days prior to Baseline
10. Use of intermittent rescue benzodiazepines (i.e., one to two doses over a 24-hour period considered one-time rescue) two or more times within the 30 days prior to Baseline

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bibbiani, Study Director — Eisai Inc.

REFERENCES:
- [Derived] Kerr WT, Brandt C, Ngo LY, Patten A, Cheng JY, Kramer L, French JA. Time to exceed pre-randomization monthly seizure count for perampanel in participants with primary generalized tonic-clonic seizures: A potential clinical end point. Epilepsia. 2022 Nov;63(11):2994-3004. doi: 10.1111/epi.17411. Epub 2022 Sep 30. PMID 36106379
- [Derived] French JA, Krauss GL, Wechsler RT, Wang XF, DiVentura B, Brandt C, Trinka E, O'Brien TJ, Laurenza A, Patten A, Bibbiani F. Perampanel for tonic-clonic seizures in idiopathic generalized epilepsy A randomized trial. Neurology. 2015 Sep 15;85(11):950-7. doi: 10.1212/WNL.0000000000001930. PMID 26296511

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 307 participants who were screened, 143 participants were screen failures and 164 participants were eligible to continue in the study but 1 participant withdrew prior to receiving treatment.
Groups:
- Placebo (Core Study): Participants received 6 tablets of perampanel matched placebo, once a day, before bedtime and with food.
- Perampanel (Core Study): Participants received 6 tablets (initially ,1 tablet of 2 mg perampanel plus 5 tablets of perampanel matched placebo) and up-titrated weekly in 2 mg increments to a target dose range of 8 mg per day maintaining the blind with administration of 6 tablets per day of either perampanel/perampanel matched placebo.
- Perampanel (Extension Phase): The Extension Phase consisted of two parts: Part A (6-week blinded Conversion Period plus a 32-week Maintenance Period) and Part B (maximum of 104-week Maintenance Period), which was followed by an additional 4-week Follow-up Period. Part A: Participants who were assigned to the perampanel arm in the Core Study continued to receive blinded perampanel once daily at the dose received during the Maintenance Period of the Core Study. During the Conversion Period, dose adjustments could be made at the investigator's discretion. Part B: Participants were unblinded to study treatment and remained on the optimal perampanel dose established during the blinded Conversion Period (Part A). Dose adjustment in 2-mg increments (upwards or downwards) was allowed at the investigator's discretion. Participants who could not tolerate a dose of 2 mg/day perampanel during the Extension Period were discontinued from the study. The maximum dose of perampanel allowed during the Extension Phase was 12 mg/day.
Period: Core Study
Arm/Group | Placebo (Core Study) | Perampanel (Core Study) | Perampanel (Extension Phase)
Started | 82 (Treated) | 81 (Treated) | 0
Completed | 72 | 68 | 0
Not Completed | 10 | 13 | 0
Not completed — Adverse Event | 5 | 9 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Participant's Choice | 2 | 3 | 0
Not completed — Inadequate therapeutic effect | 2 | 0 | 0
Period: Extension Phase
Arm/Group | Placebo (Core Study) | Perampanel (Core Study) | Perampanel (Extension Phase)
Started | 0 | 0 | 138 (Continuation into the Extension Phase was optional.)
Completed | 0 | 0 | 78
Not Completed | 0 | 0 | 60
Not completed — Adverse Event | 0 | 0 | 12
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Participant choice | 0 | 0 | 16
Not completed — Inadequate therapeutic effect | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 8
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Other | 0 | 0 | 14

BASELINE CHARACTERISTICS:
Population: The Core Study Full Analysis Set (FAS) and Extension Phase FAS included participants who were randomized to study drug, received at least 1 dose of study drug in that phase, had baseline and any postbaseline seizure frequency data during the Randomization Phase, and at least 1 observation of valid seizure diary data during treatment duration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Core Study) | Perampanel (Core Study) | Total
Number analyzed (Participants) | 82 | 81 | 163
Age, Continuous [Median (Full Range); unit: Years] | 26 [14 to 70] | 26 [12 to 58] | 26 [12 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 36 | 35 | 71

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change in Primary Generalized Tonic Clonic Seizure Frequency (PGTC) Per 28 Days During the Titration and Maintenance Periods (Combined) Relative to Baseline (Prerandomization) - (for Core Study)
Description: Seizure frequency per 28 days was derived from the information recorded in the participant diaries. PGTC seizure frequency per 28 days (as determined from participant diaries) was calculated as the number of PGTC seizures divided by the number of days in the interval and multiplied by 28. The percent change from baseline in PGTC seizure was analyzed over the Titration and Maintenance Periods combined, while baseline was defined as seizure frequency per 28 days based on all valid diary data during the Prerandomization Phase.
Time Frame: Baseline (4 or 8 weeks), Titration (4 weeks), and Maintenance (13 weeks)
Population: The Full Analysis Set included participants who were randomized to study drug, received at least 1 dose of study drug, and had any postbaseline seizure frequency data during the Randomization Phase.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo (Core Study) | Perampanel (Core Study)
Number analyzed (Participants) | 81 | 81
Percent change | -38.38 [-100 to 1546.3] | -76.47 [-100 to 184.5]
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Perampanel (Core Study); The median difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method; Test type: Superiority or Other; p = 0.0001, ANCOVA — The P-value is based on a rank analysis of covariance with treatment and pooled country as factors, and prerandomization seizure frequency as a covariate; Median Difference (Final Values) = -30.81, 95% CI 2-sided [-45.49 to -15.244]

2. Primary Outcome: 50% Responder Rate for Primary Generalized Tonic Clonic Seizure During Maintenance - LOCF - (for Core Study)
Description: A responder was a participant who experienced a 50% or greater reduction in seizure frequency per 28 days during Maintenance-last observation carried forward (LOCF) from prerandomization. The data was presented as the percentage of participants.
Time Frame: Baseline (4 or 8 weeks) and Maintenance (13 weeks)
Population: Full Analysis Set included all randomized participants who received as least 1 dose of study drug and had any postbaseline seizure frequency data. Last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (Core Study) | Perampanel (Core Study)
Number analyzed (Participants) | 81 | 81
Percentage of participants | 39.5 | 64.2
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Perampanel (Core Study); Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel — The P value is based on non-missing values and is from a Cochran-Mantel-Haenszel test stratified by pooled country

3. Primary Outcome: 50% Responder Rate in Primary Generalized Tonic-Clonic Seizure Frequency Per 28 Days Relative to the Core Study Prerandomization Phase - (for Extension Phase)
Description: Responder rate was defined as the percentage of participants who experienced a 50% or greater reduction in PGTC and total seizure frequency during treatment per 28 days relative to baseline (responder). Week 1 began on the date of first dose of the perampanel treatment regardless of whether it occurred in the Core Study or Extension Phase and continued to and included the date of the last dose of perampanel in the Extension Phase. For any given analysis window and seizure type(s), a 50% response from Core Study Prerandomization is a participant whose seizure frequency per 28 days for that seizure type(s) during that analysis window is 50% to 100% lower than his or her Core Study Prerandomization baseline seizure frequency per 28 days for that same seizure type(s). In Part B of the Extension Phase (after Visit 15), the seizure diary is only completed for days on which a seizure occurred and missing days were imputed as non-seizure days.
Time Frame: Week 1 of perampanel treatment to date of last dose of perampanel in the Extension Phase
Population: The Extension Phase FAS included participants who were eligible to participate in the Extension Phase, received at least 1 dose of study drug in this phase, and had baseline seizure frequency data and at least 1 observation of valid seizure diary data during study drug treatment duration.
Measure: Number; unit: Percentage of participants
Groups:
- Perampanel Extension Phase: The Extension Phase consisted of two parts: Part A (6-week blinded Conversion Period plus a 32-week Maintenance Period) and Part B (maximum of 104-week Maintenance Period), which was followed by an additional 4-week Follow-up Period. Part A: Participants who received placebo in the Core Study were started on blinded oral perampanel (2 mg/day) and were up-titrated weekly in 2-mg increments to the optimal dose per investigator's discretion, up to 12 mg/day perampanel maximum. Part B: Participants were unblinded to study treatment and remained on the optimal perampanel dose established during the blinded Conversion Period (Part A). Dose adjustment in 2-mg increments (upwards or downwards) was allowed at the investigator's discretion. Participants who could not tolerate a dose of 2 mg/day perampanel during the Extension Period were discontinued from the study. The maximum dose of perampanel allowed during the Extension Phase was 12 mg/day.
Arm/Group | Perampanel Extension Phase
Number analyzed (Participants) | 138
Percentage of participants
  Core Study Maintenanace Period | 55.1
  Extension Conversion Period | 74.6
  Extension Maintenance Weeks 1 to 13 | 75.9
  Extension Maintenance Weeks 14 to 26 | 78.4
  Extension Maintenance Weeks 27 to 39 | 78.1
  Extension Maintenance Weeks 40 to 52 | 79.8
  Extension Maintenance Weeks 53 to 65 | 81.8
  Extension Maintenance Weeks 66 to 78 | 76.5
  Extension Maintenance Weeks 79 to 91 | 80.3
  Extension Maintenance Weeks 92 to 104 | 91.4

4. Secondary Outcome: Median Percent Change in All Seizure Frequency Per 28 Days During the Titration and Maintenance Periods (Combined) Relative to Baseline (Prerandomization) - (for Core Study)
Description: Seizure frequency per 28 days was derived from the information recorded in the participant diaries. PGTC seizure frequency per 28 days was calculated as the number of PGTC seizures divided by the number of days in the interval and multiplied by 28. The percent change in seizure frequency relative to baseline (prerandomization) for all seizures (PGTC, myoclonic, absence and all other seizures that occur during the study) per 28 days during the Titration and Maintenance Periods combined was analyzed.
Time Frame: Baseline (4 or 8 weeks), Titration (4 weeks), and Maintenance (13 weeks)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo (Core Study) | Perampanel (Core Study)
Number analyzed (Participants) | 81 | 81
Percent Change | -22.87 [-100 to 125.7] | -43.4 [-100 to 1366.7]
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Perampanel (Core Study); The median difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method; Test type: Superiority or Other; p = 0.0018, ANCOVA — The P value is based on a rank analysis of covariance with treatment and pooled country as factors, and prerandomization seizure frequency as a covariate; Median Difference (Final Values) = -23.45, 95% CI 2-sided [-40.668 to -8.518]

5. Secondary Outcome: Median Percent Change in Primary Generalized Seizure Subtype Frequency Per 28 Days During the Titration and Maintenance Periods (Combined) Relative to Baseline (Prerandomization) - (for Core Study)
Description: Seizure frequency per 28 days was derived from the information recorded in the participant diaries. PGTC seizure frequency per 28 days was calculated as the number of PGTC seizures divided by the number of days in the interval and multiplied by 28. The percent change in seizure frequency relative to baseline (prerandomization) for primary generalized seizure subtype (myoclonic and absence) per 28 days during the Titration and Maintenance Periods combined was analyzed.
Time Frame: Baseline (4 or 8 weeks), Titration (4 weeks), and Maintenance (13 weeks)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo (Core Study) | Perampanel (Core Study)
Number analyzed (Participants) | 81 | 81
Percent Change
  Absence: number analyzed (Participants) | 33 | 27
  Absence | -7.58 [-100 to 592.4] | -41.18 [-100 to 8088.2]
  Myoclonic: number analyzed (Participants) | 23 | 24
  Myoclonic | -52.54 [-100 to 321.2] | -24.47 [-100 to 482.4]
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Perampanel (Core Study); Median Difference to Placebo for Absence Seizures; Test type: Superiority or Other; p = 0.3478, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Median Difference (Final Values) = -12.25, 95% CI 2-sided [-53.054 to 26.989] — The median difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method
Statistical Analysis 2: Comparison: Placebo (Core Study) vs Perampanel (Core Study); Median Difference to Placebo for Myoclonic Seizure; Test type: Superiority or Other; p = 0.61, ANCOVA; Mean Difference (Final Values) = 24.87, 95% CI 2-sided [-15.338 to 59.938]

6. Secondary Outcome: 50% Responder Rate for All Seizures During Maintenance-LOCF - (for Core Study)
Description: All seizures included PGTC, myoclonic, absence and all other seizures that occur during the study. A responder was a participant who experienced a 50% or greater reduction in seizure frequency per 28 days during Maintenance- LOCF from prerandomization. The data was presented as percentage of participants.
Time Frame: Baseline (4 or 8 weeks) and Maintenance (13 weeks)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (Core Study) | Perampanel (Core Study)
Number analyzed (Participants) | 81 | 81
Percentage of participants | 34.6 | 45.7
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Perampanel (Core Study); Test type: Superiority or Other; p = 0.1826, Cochran-Mantel-Haenszel — The P value is based on non-missing values and is from a Cochran-Mantel-Haenszel test stratified by pooled country

7. Secondary Outcome: 50% Responder Rate for Primary Generalized Seizure Subtype During Maintenance Period - LOCF - (for Core Study)
Description: Primary generalized seizure subtype included absence and myoclonic seizures. A responder was a participant who experienced a 50% or greater reduction in seizure frequency per 28 days during Maintenance - (LOCF) from prerandomization. The data was presented as the percentage of participants.
Time Frame: Baseline (4 or 8 weeks) and Maintenance (13 weeks)
Population: Only a subset of participants in the Full Analysis Set who experienced these seizure types during the Prerandomization Phase of the study were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (Core Study) | Perampanel (Core Study)
Number analyzed (Participants) | 81 | 81
Percentage of participants
  Absence: number analyzed (Participants) | 33 | 27
  Absence | 39.4 | 48.1
  Myoclonic: number analyzed (Participants) | 23 | 24
  Myoclonic | 60.9 | 41.7
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Perampanel (Core Study); P Value Compared to Placebo for Absence Seizures; Test type: Superiority or Other; p = 0.4653, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo (Core Study) vs Perampanel (Core Study); P Value Compared to Placebo for Myoclonic Seizures; Test type: Superiority or Other; p = 0.3694, Cochran-Mantel-Haenszel

8. Secondary Outcome: Percent Change From Core Study Prerandomization Phase in Primary Generalized Tonic-Clonic (PGTC) Seizure Frequency Per 28 Days - (for Extension Phase)
Description: Week 1 began on the date of first dose of the perampanel treatment regardless of whether it occurred in the Core Study or Extension Phase and continued to and included the date of the last dose of perampanel in the Extension Phase. For any given analysis window and seizure type(s), a 50% responder from Core Study Randomization is a participant whose seizure frequency per 28 days for that seizure type(s) during that analysis window is 50% to 100% lower than his or her Core Study Prerandomization baseline seizure frequency per 28 days for that same seizure type(s). In Part B of the Extension Phase (after Visit 15), the seizure diary is only completed for days on which a seizure occurred and missing days were imputed as non-seizure days.
Time Frame: Date of first dose of study drug to date of last dose of study drug in the Extension Phase
Population: Full analysis set included all participants who were eligible to participate in the Extension Phase, received at least 1 dose of perampanel in this phase, and had baseline seizure frequency data and at least 1 observation of valid seizure diary data during the perampanel treatment duration.
Measure: Median (Full Range); unit: Percent change in PGTC seizure frequency
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 138
Percent change in PGTC seizure frequency
  Core Study Titration Period | -57.72 [-100.0 to 500.0]
  Core Study Maintenance Period | -57.40 [-100.0 to 2011.6]
  Extension Phase Conversion Period | -100.00 [-100.0 to 166.7]
  Extension Phase Maintenance Period, Weeks 1 to 13: number analyzed (Participants) | 133
  Extension Phase Maintenance Period, Weeks 1 to 13 | -84.62 [-100.0 to 594.5]
  Extension Phase Maintenance Period, Weeks 14 to 26: number analyzed (Participants) | 125
  Extension Phase Maintenance Period, Weeks 14 to 26 | -86.81 [-100.0 to 186.2]
  Extension Phase Maintenance Period, Weeks 27 to 39: number analyzed (Participants) | 114
  Extension Phase Maintenance Period, Weeks 27 to 39 | -86.62 [-100.0 to 250.8]
  Extension Phase Maintenance Period, Weeks 40 to 52: number analyzed (Participants) | 104
  Extension Phase Maintenance Period, Weeks 40 to 52 | -100.00 [-100.0 to 146.2]
  Extension Phase Maintenance Period, Weeks 53 to 65: number analyzed (Participants) | 99
  Extension Phase Maintenance Period, Weeks 53 to 65 | -100.00 [-100.0 to 150.5]
  Extension Phase Maintenance Period, Weeks 66 to 78: number analyzed (Participants) | 68
  Extension Phase Maintenance Period, Weeks 66 to 78 | -100.00 [-100.0 to 108.8]
  Extension Phase Maintenance, Weeks 79 to 91: number analyzed (Participants) | 61
  Extension Phase Maintenance, Weeks 79 to 91 | -100.00 [-100.0 to 140.1]
  Extension Phase Maintenance, Weeks 92 to 104: number analyzed (Participants) | 35
  Extension Phase Maintenance, Weeks 92 to 104 | -100.00 [-100.0 to 171.4]

9. Secondary Outcome: Summary of Percent Change From Pre-Perampanel Baseline in Seizure Frequency Per 28 Days - (for Extension Phase)
Description: Efficacy assessments included seizure counts from participant diaries. The percent change in seizure frequency was assessed during the perampanel treatment duration, with the pre-perampanel baseline being used for evaluating the change. The pre-perampanel baseline was defined as follows: 1) for all participants who had been assigned to placebo treatment in the Core Study, the pre-perampanel baseline was computed from all valid seizure diary data during the Core Study, and 2) for participants who had been assigned to perampanel in the Core Study, the pre-perampanel baseline was computed from all valid seizure diary data during the Prerandomization Phase plus the 4 weeks prior to the Prerandomization Phase of the Core Study. The perampanel treatment duration consisted of: 1) the Randomization Phase of the Core Study plus the Extension Phase for participants assigned to perampanel in the Core Study, and 2) the Extension Phase for participants assigned to placebo in the Core Study.
Time Frame: Weeks: 1 to 13, 14 to 26, 27 to 39, 40 to 52, 53 to 65, 66 to 78, 79 to 91, 92 to 104, 105 to 117, 118 to 130, 131 to 143, greater than or equal to 144
Population: Full Analysis Set, which comprised all participants who were eligible to participate in the Extension Phase, received at least 1 dose of perampanel in this phase, and had baseline seizure frequency data and at least 1 observation of valid seizure diary data during the perampanel treatment duration.
Measure: Median (Full Range); unit: Percent change in seizure frequency
Groups:
- PGTC Seizures: The median percent change from the Pre-perampanel baseline in PGTC seizure frequency per 28 days by 13-week intervals through greater than or equal to Week 144.
- All Seizures: The median percent change from the Pre-perampanel baseline in the seizure frequency per 28 days of all seizures by 13-week intervals through greater than or equal to Week 144.
Arm/Group | PGTC Seizures | All Seizures
Number analyzed (Participants) | 138 | 138
Percent change in seizure frequency
  Weeks 1 to 13 | -77.45 [-100.0 to 676.9] | -56.54 [-100.0 to 1130.8]
  Weeks 14 to 26: number analyzed (Participants) | 133 | 133
  Weeks 14 to 26 | -74.21 [-100.0 to 191.7] | -63.53 [-100.0 to 1253.8]
  Weeks 27 to 39: number analyzed (Participants) | 125 | 125
  Weeks 27 to 39 | -84.62 [-100.0 to 264.4] | -79.49 [-100.0 to 1100.0]
  Weeks 40 to 52: number analyzed (Participants) | 118 | 118
  Weeks 40 to 52 | -89.65 [-100.0 to 171.9] | -83.38 [-100.0 to 855.6]
  Weeks 53 to 65: number analyzed (Participants) | 109 | 109
  Weeks 53 to 65 | -92.45 [-100.0 to 49.6] | -83.33 [-100.0 to 54.8]
  Weeks 66 to 78: number analyzed (Participants) | 90 | 90
  Weeks 66 to 78 | -100.00 [-100.0 to 92.3] | -88.71 [-100.0 to 100.5]
  Weeks 79 to 91: number analyzed (Participants) | 80 | 80
  Weeks 79 to 91 | -100.00 [-100.0 to 700.0] | -90.28 [-100.0 to 700.0]
  Weeks 92 to 104: number analyzed (Participants) | 52 | 52
  Weeks 92 to 104 | -100.00 [-100.0 to 171.4] | -98.96 [-100.0 to 394.4]
  Weeks 105 to 117: number analyzed (Participants) | 41 | 41
  Weeks 105 to 117 | -100.00 [-100.0 to 118.2] | -96.42 [-100.0 to 118.2]
  Weeks 118 to 130: number analyzed (Participants) | 27 | 27
  Weeks 118 to 130 | -100.00 [-100.0 to -8.5] | -96.58 [-100.0 to 27.8]
  Weeks 131 to 143: number analyzed (Participants) | 19 | 19
  Weeks 131 to 143 | -100.00 [-100.0 to 20.1] | -91.70 [-100.0 to -52.7]
  Weeks greater than or equal to 144: number analyzed (Participants) | 9 | 9
  Weeks greater than or equal to 144 | -100.00 [-100.0 to -71.5] | -82.09 [-100.0 to -31.3]

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events as a Measure of Safety and Tolerability of Perampanel in Subjects With Inadequately Controlled PGTC Seizures - (for Core Study)
Description: An Adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered an investigational product. A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening (i.e., the subject was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect (in the child of a subject who was exposed to the study drug). In this study, treatment emergent adverse events (TEAEs) (defined as an AE that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) were assessed.
Time Frame: For each participant, from the first treatment dose till 30 days after the last dose or up to 21 weeks for core study and 142 weeks for extension phase.
Population: The Safety Analysis Set included participants who were randomized to study drug, received at least 1 dose of study drug, and had at least 1 postbaseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Core Study) | Perampanel (Core Study)
Number analyzed (Participants) | 82 | 81
Participants
  Treatment emergent adverse events | 59 | 67
  Treatment emergent serious adverse events | 7 | 6

ADVERSE EVENTS:
Time Frame: From the date of first dose of perampanel up to 30 days after the last dose, or up to approximately 163 weeks total.
Description: Treatment-emergent Adverse Events (TEAEs) included AEs that occurred from the first dose of perampanel (in Core Study or Extension Phase) to 30 days after the last dose of perampanel, or that were present before the first day of perampanel administration but worsened in severity during the study. TEAEs are reported in the Safety Section.
Arm/Group | Placebo (Core Study) | Perampanel (Core Study) | Perampanel (Extension Phase)
Serious Adverse Events (participants affected / at risk) | 7/82 | 6/81 | 18/138
Other Adverse Events (participants affected / at risk) | 56/82 | 67/81 | 106/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Core Study) (N=82) | Perampanel (Core Study) (N=81) | Perampanel (Extension Phase) (N=138)
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Drowning (General disorders) | 0 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 1 | 3
Grand Mal Convulsion (Nervous system disorders) | 1 | 0 | 1
Status Epilepticus (Nervous system disorders) | 1 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sedation (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Psychiatric symptom (Psychiatric disorders) | 0 | 0 | 1
Psychogenic seizure (Psychiatric disorders) | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Core Study) (N=82) | Perampanel (Core Study) (N=81) | Perampanel (Extension Phase) (N=138)
Vertigo (Ear and labyrinth disorders) | 2 | 7 | 15
Abdominal Pain (Gastrointestinal disorders) | 1 | 4 | 8
Nausea (Gastrointestinal disorders) | 3 | 5 | 11
Vomiting (Gastrointestinal disorders) | 2 | 7 | 9
Fatigue (General disorders) | 5 | 12 | 14
Irritability (General disorders) | 2 | 9 | 19
Nasopharyngitis (Infections and infestations) | 7 | 7 | 20
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 4 | 18
Contusion (Injury, poisoning and procedural complications) | 3 | 5 | 12
Weight Increased (Investigations) | 3 | 6 | 13
Dizziness (Nervous system disorders) | 5 | 26 | 53
Headache (Nervous system disorders) | 8 | 10 | 17
Somnolence (Nervous system disorders) | 3 | 9 | 18
Anxiety (Psychiatric disorders) | 3 | 4 | 7
Insomnia (Psychiatric disorders) | 4 | 3 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other